CLINICAL TRIAL: NCT06245265
Title: Evaluation of the Effect of Non-Surgical Periodontal Therapy on Serum and Salivary Biomarker Levels in Individuals With Rheumatoid Arthritis
Brief Title: The Effect of Non-Surgical Periodontal Therapy on Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Burcu KARADUMAN, Professor, Biruni University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-KAEK-80-23-02
Record Dates: First submitted 2024-01-26; First posted 2024-02-07 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2024-02

CONDITIONS: Periodontitis; Rheumatoid Arthritis
Keywords: Periodontititis; Rheumatoid arthritis; Cytokine
MeSH Terms: conditions — Periodontitis; Arthritis, Rheumatoid | interventions — Enzyme-Linked Immunosorbent Assay

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Clinical Healthy (Experimental): Clinical measurements (Plaque index, probing depth, gingival recession, clinical attachment level, bleeding on probing) salivary sample and serum will be taken from all individuals at the beginning of the study. ANGPTL-4 levels will be examined to evaluate before and after treatment in periodontal health and periodontitis. A pre-treatment saliva sample and serum will be collected from the clinically healthy group.
  Interventions: Other: ELISA (Enzyme-Linked ImmunoSorbent Assay)
- Periodontitis (Experimental): Non-surgical periodontal treatment will be applied to individuals with periodontitis, clinical measurements, saliva collection and serum will be repeated 12 weeks after the treatment. ANGPTL-4 analysis will be performed by ELISA in saliva and serum of individuals. ANGPTL-4 levels will be examined to evaluate before and after treatment in periodontal health and periodontitis. Clinical measurements (Plaque index, probing depth, gingival recession, clinical attachment level, bleeding on probing) and salivary sample will be taken from all individuals at the beginning of the study.
  Interventions: Other: ELISA (Enzyme-Linked ImmunoSorbent Assay)
- Periodontitis with rheumatoid arthritis (Experimental): Non-surgical periodontal treatment will be applied to individuals with periodontitis, clinical measurements, saliva collection and serum will be repeated 12 weeks after the treatment. ANGPTL-4 analysis will be performed by ELISA in saliva and serum of individuals. ANGPTL-4 levels will be examined to evaluate before and after treatment in periodontitis with rheumatoid arthritis. Clinical measurements (Plaque index, probing depth, gingival recession, clinical attachment level, bleeding on probing) and salivary sample will be taken from all individuals at the beginning of the study.
  Interventions: Other: ELISA (Enzyme-Linked ImmunoSorbent Assay)
- Healthy individuals with RA (Experimental): Clinical measurements (Plaque index, probing depth, gingival recession, clinical attachment level, bleeding on probing) salivary sample and serum fluid will be taken from all individuals at the beginning of the study. ANGPTL-4 levels will be examined to evaluate before and after treatment in periodontal health and periodontitis. A pre-treatment saliva sample and serum will be collected from the healthy individuals with RA group.
  Interventions: Other: ELISA (Enzyme-Linked ImmunoSorbent Assay)

INTERVENTIONS:
Other: ELISA (Enzyme-Linked ImmunoSorbent Assay) — In this study, 15 periodontitis patients with RA, 15 healthy individuals with RA, 15 systemic healthy periodontitis patients and 15 systemic periodontally healthy individuals will be included. ANGPTL-4 biomarker and other biomarkers (MMP-13, TNF-α, IL-6) that have not been previously analysed in the serum and saliva of both RA and periodontitis patients will be evaluated before and 3 months after COPT. Clinical parameters (Plaque index, probing depth, gingival recession, clinical attachment level, bleeding on probing), biochemical evaluations of serum, saliva and gingival samples will be performed and correlated with clinical parameters at baseline and 3 months after COPT in all individuals with periodontitis included in the study.

SUMMARY:
Periodontitis is a common chronic inflammatory disease characterised by the destruction of the soft and hard tissues supporting the tooth, including alveolar bone, periodontal ligament and cementum. Periodontitis has been associated with different host characteristics such as diabetes or neutrophil disorders and environmental factors such as smoking, alcohol consumption and stress. On the other hand, periodontal bacterial infection triggers a systemic immune response that is associated with an increased risk of different disorders such as bacterial pneumonia, cardiovascular disease and autoimmune diseases. Rheumatoid arthritis (RA) is a severe chronic autoimmune disease of unknown etiology, characterised by symmetrical, erosive synovitis of the joints, sometimes with multisystem organ involvement, joint destruction and excessive bone loss. Although the etiology of RA is unknown, it is thought to occur in individuals with genetic predisposition as a result of exposure to various environmental factors. RA and periodontitis are chronic destructive inflammatory diseases with common genetic and environmental risk factors, pathogenesis mechanisms and complex multifactorial pathological processes. Several studies suggest that periodontitis, a common inflammatory disease of the periodontium surrounding the teeth and triggered by bacteria in the mouth, is associated with RA and may initiate and worsen inflammation in RA. Non-surgical periodontal treatment (COPT), which is considered the gold standard in the treatment of periodontitis with hand instruments and ultrasonic instruments, has been shown to provide significant improvements in the clinical outcomes of periodontitis patients with RA. COPT is performed to stop the progression of periodontal diseases. Considering the studies supporting the bidirectional relationship between periodontitis and RA, it is thought that COPT may affect the clinical and biochemical values of RA. Based on these points, the aim of our study was to investigate the relationship between serum and salivary ANGPTL-4, MMP-13, TNF-α and IL-6 levels and periodontal disease in individuals with RA and to evaluate the effects of COPT on RA disease severity in vivo.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 18-65,
* Having at least 8 teeth excluding wisdom teeth,
* No periodontal treatment in the last 3 months,
* Not having used antibiotics in the last 3 months,
* Not being pregnant or breastfeeding,
* The individuals to be included in the control group should not have any systemic disease that may change the periodontal status, and the individuals to be included in the experimental group should not have any systemic disease that may affect periodontal health except RA.

Exclusion Criteria:

* Under 18 years of age and over 65 years of age,
* Having less than 8 teeth,
* Having undergone periodontal treatment in the last 3 months,
* Having used antibiotics in the last 3 months,
* Being pregnant or breastfeeding,
* Individuals to be included in the control group should have any systemic disease that may change the periodontal status, and individuals to be included in the test group should have any systemic disease that may affect periodontal health except RA.
* Abnormal body mass index (more than 29.9 kg/m2).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Examination of ANGPTL-4 levels of periodontal disease and rheumatoid arthritis | up to 1 year
  Examination of ANGPTL-4 levels, which are stated to be associated with periodontal disease, in serum and saliva samples obtained from individuals with periodontitis and periodontitis individuals with RA.

SECONDARY OUTCOMES:
Evaluation of the effect of non-surgical periodontal treatment on changes in ANGPTL-4 level. | up to 1 year
  Evaluation of the effect of non-surgical periodontal treatment on changes in ANGPTL-4 level.

OTHER OUTCOMES:
Comparison biomarkers of study groups. | up to 1 year
  Comparison of serum and saliva samples taken before treatment in individuals with periodontitis and periodontitis individuals with RA in terms of ANGPTL-4 levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No